CLINICAL TRIAL: NCT02603289
Title: One Week Aligner Evaluation
Status: Completed | Type: Observational
Sponsor: Align Technology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP-300313-00
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion | interventions — Orthodontic Appliances, Removable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Teen: < 17 years of age
  Interventions: Device: Invisalign
- Adult: 17 years of age or older
  Interventions: Device: Invisalign
- Adult with Primer Aligners: 17 years of age or older This group will get Primer Aligners
  Interventions: Device: Invisalign

INTERVENTIONS:
Device: Invisalign

SUMMARY:
The purpose of this study is to demonstrate that changing aligners weekly provides similar results to changing aligners every two weeks.

DETAILED DESCRIPTION:
The Invisalign® System consists of a series of clear plastic aligners that are intended to replace conventional wire and bracket technology for many orthodontic cases. Each custom manufactured aligner exerts gentle, continuous forces to move teeth incrementally from their original state to a final, treated state. The aligners are designed to optimally move each tooth at a speed that follows physiologic principles. The purpose of this study is to demonstrate that changing aligners weekly provides similar results to changing aligners every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have fully erupted dentition except for 2nd and 3rd molars
* For Teen treatment group, subjects ages <17 years of age
* For Adult treatment group, subjects ≥17 years of age

Exclusion Criteria:

* Subject has undergone any accelerated orthodontic treatment prior to or during treatment as part of this study
* Subject with active caries
* Subject with periodontal disease
* Subject with TMD symptoms
* Subject has known allergy to latex or plastic
* Subjects who are pregnant or will become pregnant during treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Invisalign patients from selected pool of investigators
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Planned to Final Tooth Position | Through study completion, an average of 2 years
  Test vs Historical Control Group

SECONDARY OUTCOMES:
Treatment time | Through study completion, an average of 2 years
  Length of treatment
Subject Quality of Life | Through study completion, an average of 2 years
  Assessment of QoL

CONTACTS AND LOCATIONS:
Locations (24):
- United States (23):
  - Dr. Thomas Marcel, Livermore, California
  - Dr. Mary Cooke, Napa, California
  - Dr. Bella Shen Garnett, San Francisco, California
  - Align Technology, Inc., San Jose, California
  - Dr. Robery Van den Berg, San Ramon, California
  - Dr. Anil Idiculla, Lone Tree, Colorado
  - Dr. Ryan Caudill, Merritt Island, Florida
  - Dr. Sean Holliday, Pearl City, Hawaii
  - Dr. Jeff Mastroianni, Glen Carbon, Illinois
  - Dr. Mark Perelmuter, Louisville, Kentucky
  - Dr. James Crouse, Salisbury, Maryland
  - Dr. Zvi Kennet, Macomb, Michigan
  - Dr. Thomas Everett, Burnsville, Minnesota
  - Dr. Justin Wild, Eden Prairie, Minnesota
  - Dr. Regina Blevins, Inver Grove Heights, Minnesota
  - Dr. William Kottemann, Maple Grove, Minnesota
  - Dr. Vincent D'Ascoli, Carson City, Nevada
  - Dr. David Chenin, Henderson, Nevada
  - Dr. Carlyn Phucas, Marlton, New Jersey
  - Dr. David Paquette, Mooresville, North Carolina
  - Dr. William Gierie, Wilmington, North Carolina
  - Dr. Brian Amy, Oklahoma City, Oklahoma
  - Dr. Clark Colville, Seguin, Texas
- Dr. Bart Iwasiuk, Brampton, Ontario, Canada